CLINICAL TRIAL: NCT05735951
Title: Open Label, Phase I Study to Assess and Compare the Pharmacokinetic Parameters After Multiple Oral Administration of Stiripentol 1000 mg in Renal Impaired Patients and Matching Controls With Normal Renal Function
Brief Title: Pharmacokinetic Parameters of Stiripentol in Renal Impaired Patients and Matching Controls With Normal Renal Function
Acronym: STP237
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JADE
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Chronic Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Mild renally impaired patients (Experimental): Mild renally impaired patients
  Interventions: Drug: STIRIPENTOL oral administration
- Moderate renally impaired patients (Experimental): Moderate renally impaired patients
  Interventions: Drug: STIRIPENTOL oral administration
- Severe renally impaired patients (Experimental): Severe renally impaired patients
  Interventions: Drug: STIRIPENTOL oral administration
- Matching controls (Experimental): Matching volunteer without renal impairement
  Interventions: Drug: STIRIPENTOL oral administration

INTERVENTIONS:
Drug: STIRIPENTOL oral administration — Oral administration of:
  * Days 1 and 2: 1000 mg of stiripentol (single dose at the end of breakfast),
  * Day 3 to Day 14: 1000 mg of stiripentol bis in die (BID) (approximately 12 hours apart, at the end of breakfast and at the end of dinner),
  * Day 15: 1000 mg of stiripentol (single dose at the end of breakfast).
  Other Names: Multiple oral administration of stiripentol 1000 mg bis in die (BID)

SUMMARY:
The purpose of this study is to determine whether the pharmacokinetics (PK) of stiripentol and of its relevant metabolites would be altered in subjects with renal impairment compared with normal controls in order to assess the need of dose adjustment in the renal impaired population. This study will include subjects with mild, moderate and severe renal impairment.

DETAILED DESCRIPTION:
The pharmacokinetic studies conducted with stiripentol in humans evidenced that at steady state after multiple administration, up to 54.1%. of the stiripentol dose was excreted unchanged in hydrolyzed urine over the 24 h interval. Stiripentol is extensively metabolized by the liver; around 20 metabolites have been detected in urine, but the fraction of dose excreted as unchanged stiripentol is much less than one percent. At steady state, stiripentol and its metabolites in urine accounted collectively for 90% of the oral dose.

The risk of a clinically relevant increase in exposure in renal impairment is expected to be largest for drugs that are primarily renally eliminated, according to the European Medicines Agency (EMA) guideline on the evaluation of the pharmacokinetics of medicinal products in patients with decreased renal function and the draft Food and Drug Administration's (FDA) guidance for industry "Pharmacokinetics in Patients with Impaired Renal Function - Study Design, Data Analysis, and Impact on Dosing and Labeling". But since the literature shows that impaired renal function can alter some drug metabolism and transport pathways in the liver and gut a dedicated renal impairment study with a full pharmacokinetics (PK) design is recommended.

Therefore, the purpose of this study is to determine whether the pharmacokinetics (PK) of stiripentol and of its relevant metabolites would be altered in subjects with renal impairment compared with normal controls in order to assess the need of dose adjustment in the renal impaired population. This study will include subjects with mild, moderate and severe renal impairment.

Data from subjects with renal impairment will be compared to matched controls with normal renal function. Both groups should be similar with respect to sex, age, BMI and ethnicity. This approach is consistent with recommendations of the EMA guideline and FDA guidance for pharmacokinetics (PK) in patients with renal function as the control group in this study should be representative of the typical patient population for the drug under study, considering the patients' renal function and other factors known to affect the drug's pharmacokinetics (PK).

Plasma protein binding is often altered in patients with impaired renal function. Stiripentol is strongly bound (>99%) to plasma proteins. Therefore, the EMA guideline and FDA guidance recommend the measurement of unbound drug concentrations. Therefore, the fraction of unbound stiripentol will be determined using two samples taken pre-dose and 3 h post-dose on Day 15 from each subject on-study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects

Subjects/patients will be required to satisfy all the following inclusion criteria to be included in the study:

1. Male or female subjects, aged 18 to 80 years inclusive,
2. Females participating in this study must be of non-childbearing potential or using highly effective contraception for the full duration of the study and for 1 month after the end of treatment,
3. Negative serum pregnancy test at screening and urinary pregnancy test at Day -1 (if applicable),
4. A negative antigen test for Coronavirus Disease 19 (COVID 19),
5. Normal hepatic function (AST < 3xULN (Upper limit normal), ALT (Alanine aminotransferase); <1.5 ULN; bilirubin),
6. Non-smoker subject or smoker of not more than 5 cigarettes a day,
7. Signing a written informed consent in their native language prior to selection,

Additional inclusion criteria for renally impaired patients

Patients with renal impairment will be required to satisfy all the following inclusion criteria to be included in the study:

1. Documented renal impairment indicated by reduced RF at least 12 months of screening or longer,
2. Stable renal function (eGFR) as evidenced by ≤ 30% difference in two evaluations of Renal function (RF) on two separate occasions separated by at least 28 days with one measurement being the value at screening,
3. Renal impairment within the following ranges (using the Modification of Diet in Renal Disease-4 (MDRD4) equation) at screening:

   1. mild renal impairment with eGFR ≥ 60 to < 90 mL/min/1.73 m²,
   2. moderate renal impairment with eGFR ≥ 30 to < 60 mL/min/1.73 m²,
   3. severe renal impairment with eGFR < 30 mL/min/1.73 m² and not on dialysis,
4. Supine blood pressure (BP) ≤ 180/104 mmHg,
5. Heart rate between 50-100 bpm, DBP between 40-100 mmHg and SBP between 90-170 mmHg extremities excluded,
6. Normal or non-clinically significant finding in ECG recording on a 10 min resting 12-lead ECG at the screening visit (left ventricular hypertrophy related with hypertension, will be allowed):

   * HR [50-100 bpm],
   * 110 ms ≤ interval between P and R waves (PR) < 220 ms,
   * Interval between Q and S waves (QRS) < 120 ms,
   * Fridericia corrected interval between Q and T waves (QTcF) ≤ 450 ms, 470 ms for female,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCS by the Investigator,
7. Body Mass Index (BMI) between 18 and 35 kg/m² inclusive.

Additional inclusion criteria for matching controls

Matching controls will be required to satisfy all the following inclusion criteria to be included in the study:

1. Considered as healthy after a comprehensive clinical assessment (detailed medical history and complete physical examination),
2. eGFR ≥ 90 mL/min/1.73 m²,
3. No proteinuria (i.e., no trace or positive dipstick results),
4. BMI between 18 and 35 kg/m2 inclusive and body weight,
5. Normal BP and heart rate (HR) at the screening visit after 5 min in supine position:

   * 90 mmHg ≤ Systolic Blood Pressure (SBP) ≤ 145 mmHg, for elderly subjects (> 60 years) an upper limit of 150 mmHg,
   * 45 mmHg ≤ Diastolic Blood Pressure (DBP) ≤ 90 mmHg, for elderly subjects (> 60 years) an upper limit of 95 mmHg,
   * 50 bpm ≤ HR ≤ 100 bpm,
   * Or value outside these limits but considered not clinically significant (NCS) by the Investigator,
6. Normal ECG recording on a 10 min resting 12-lead ECG at the screening visit:

   * HR [50-100 bpm],
   * 110 ≤ interval between P and R waves (PR) < 220 ms,
   * Interval between Q and S waves (QRS) < 120 ms,
   * Fridericia corrected interval between Q and T waves (QTcF) ≤ 450 ms, 470 ms for female,
   * No sign of any trouble of sinusal automatism,
   * Or considered NCS by the Investigator,
7. Laboratory parameters within the normal range or considered NCS by the Investigator of the laboratory (hematological, blood chemistry tests, urinalysis). Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator,
8. Normal dietary habits,
9. Matched to at least 1 renally impaired patient by ethnic group, sex, age (+/- 10 years) and BMI (+/-20%).

Exclusion Criteria:

Non-inclusion criteria for all subjects

All the subjects/patients included in the study must not meet any of the following non-inclusion criteria:

1. Unsuitable veins for repeated venipuncture,
2. Positive Hepatitis B surface (HBsAg) antigen or positive Hepatitis C Virus (HCV), or positive results for Human Immunodeficiency Virus (HIV)-1 or 2 tests,
3. History or presence of drug or alcohol abuse (alcohol consumption >40 grams/day),
4. Subject/Patient who, in the judgment of the Investigator, is likely to be non-compliant or uncooperative during the study, or unable to cooperate because of a language problem, poor mental development,
5. Subject/Patient who cannot be contacted in case of emergency,
6. History or presence of allergy or unusual reactions to some drugs or anesthetics or known hypersensitivity to the investigation product or its excipients (including lactose intolerance), test material or related compound,
7. Who receive a medication known to affect both cyochromes (CYP) CYP1A2, CYP3A4, and CYP2C19, such as rifampin, within 1 month prior to the first dose administration. Concomitant use of medications known to strongly affect either CYP1A2, CYP3A4, or CYP2C19, such as phenytoin, phenobarbital or carbamazepine, should be avoided within 1 month prior to the first dose administration.
8. Subject/Patient who is in the exclusion period of a previous study,
9. Administrative or legal supervision,
10. Blood donation (including in the frame of a clinical trial) within 2 months before administration,
11. Subject/Patient who is pregnant, in labour or breastfeeding. Subject/Patient should not be enrolled if she plans to become pregnant during the time of study participation,
12. Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day),
13. Positive COVID 19 antigen test, or COVID-19 vaccination within 14 days of the first dosing.
14. The consumption of grapefruit/grapefruits production, Sevilla oranges, or any poppy seeds, are not allowed from 7 days prior to the first study drug administration,
15. Evidence or history of clinically significant uncontrolled hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, metabolic, systemic, infectious, or allergic disease (including drug hypersensitivity or allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing). However, investigator will have the possibility to judge whether a subject could be included with uncontrolled disease (e.g. in case of non-treated dyslipidemia),
16. General anesthesia within 3 months before administration,
17. Major surgery within 28 days prior to inclusion or major surgery planned during the next 6 months,
18. Inability to abstain from intensive muscular effort,
19. Inability or difficulty swallowing whole capsules,

Additional non-inclusion criteria for renal impaired patients

Patients with renal impairment included in the study must not meet any of the following non-inclusion criteria:

1. History of renal transplant,
2. The patient has evidence of an unstable clinically important medical condition other than impaired renal function,
3. The patient has an acute exacerbation or unstable renal function, as indicated by worsening of clinical and/or laboratory signs of renal impairment, within the 4 weeks before study drug administration,
4. Patients undergoing any method of dialysis or hemofiltration,
5. Disorders or surgery of the gastrointestinal tract which may interfere with drug absorption or may otherwise influence the pharmacokinetics (PK) of the investigational medicinal product (IMP) (e.g., inflammatory bowel disease, resections of the small or large intestine, etc.),
6. History of febrile illness within 5 days prior to dosing,
7. Evidence of clinically significant liver disease or liver damage (e.g., hepatitis B or C, autoimmune hepatitis, primary biliary cirrhosis, non-alcoholic fatty liver disease, elevated aspartate aminotransferase (AST) or ALT that is considered clinically significant by the Investigator, etc.),
8. Patient with a change in current treatments during the last month or receiving any drug known to be potent CYP1A2, CYP3A4 and CYP2C19 inducers, such as rifampin.

   Additional non-inclusion criteria for matching controls Matching controls with normal renal function included in the study must not meet any of the following noninclusion criteria:
9. Any history or presence of renal disease,
10. Frequent headaches (> twice a month) and / or migraines, recurrent nausea and / or vomiting,
11. Symptomatic hypotension whatever the decrease of blood pressure or asymptomatic postural hypotension defined by a decrease in SBP (≥20 mmHg) or DBP (≥10 mmHg) within 2 min when changing from the supine to the standing position, Intake of any medication (except paracetamol, hormonal contraceptives and hormone replacement therapy for post-menopausal women), including over the counter (OTC) medications and herbal products, that could affect the outcome of the study is prohibited within 2 weeks prior to the first drug administration or less than 5 times the t1/2 of that drug, whichever is the longer, or participant receiving any drug known to interfere with CYP enzymes within 1 month prior to the first dose administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve | Steady state at Day15
  Area under the plasma concentration versus time curve: AUC0-12 (corresponding to AUC0-tau), in order to assess the need of dose adjustment in the renal impaired population.
Peak Plasma Concentration | Steady state at Day15
  Peak Plasma Concentration: Cmax in order to assess the need of dose adjustment in the renal impaired population.

SECONDARY OUTCOMES:
Peak Plasma Concentration, for stiripentol in plasma | Day 1 and Day 15 when applicable
  Peak Plasma Concentration : Cmax on Day 1
The area under the concentration-time curve from time zero (pre-dose) to 12 h post-dose, for stiripentol in plasma | Day 1 and Day 15 when applicable
  The area under the concentration-time curve from time zero (pre-dose) to 12 h post-dose: AUC0-12 corresponds to AUC0-tau on Day 15): AUC0-12 on Day 1
The time at which Cmax is apparent, for stiripentol in plasma | Day 1 and Day 15 when applicable
  The time at which Cmax is apparent: tmax
The area under the concentration-time curve from time zero (pre-dose) to 24 h post-dose, for stiripentol in plasma | Day 1 and Day 15 when applicable
  The area under the concentration-time curve from time zero (pre-dose) to 24 h post-dose: AUC0-24,
The area under the concentration-time from time zero (pre-dose) to the time of last quantifiable concentration, for stiripentol in plasma | Day 1 and Day 15 when applicable
  The area under the concentration-time from time zero (pre-dose) to the time of last quantifiable concentration: AUC0-t
The apparent terminal elimination half-life, for stiripentol in plasma | Day 1 and Day 15 when applicable
  The apparent terminal elimination half-life t1/2
Apparent total clearance at steady-state, for stiripentol in plasma | Day 1 and Day 15 when applicable
  Apparent total clearance at steady-state: CLss/F
Fraction unbound (stiripentol) in plasma defined as unbound concentration/total concentration (on Day 15 only), for stiripentol in plasma | Day 1 and Day 15 when applicable
  Fraction unbound (stiripentol) in plasma defined as unbound concentration/total concentration (on Day 15 only) : Fu
Pre-morning dose concentration, for stiripentol in plasma | Day 1 and Day 15 when applicable
  Pre-morning dose concentration : Cmin
Accumulation ratio evaluated, for stiripentol in plasma | Day 1 and Day 15 when applicable
  Accumulation ratio evaluated: Racc
Total amount excreted over the time interval between 0 and 12 h, for stiripentol in urine | Day 1 and Day 15 when applicable
  Total amount excreted over the time interval between 0 and 12 h : Ae0-12
Total amount excreted over the total time interval of urine collection i.e. ]0 - 24] h, for stiripentol in urine | Day 1 and Day 15 when applicable
  Total amount excreted over the total time interval of urine collection i.e. ]0 - 24] h : Ae0-24
The fraction of the dose excreted in urine over the total time interval of urine collection i.e. ]0 - 24] h, for stiripentol in urine | Day 1 and Day 15 when applicable
  The fraction of the dose excreted in urine over the total time interval of urine collection i.e. ]0 - 24] h : fe0-24
The renal clearance, for stiripentol in urine | Day 1 and Day 15 when applicable
  The renal clearance : CLr
Peak Plasma Concentration, for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  Peak Plasma Concentration : Cmax
The time at which Cmax is apparent, for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  Peak Plasma Concentration : Cmax
The area under the concentration-time curve from time zero (pre-dose) to 12 h post-dose: AUC0-12 corresponds to AUC0-tau on Day 15), for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  The area under the concentration-time curve from time zero (pre-dose) to 12 h post-dose: AUC0-12 corresponds to AUC0-tau on Day 15) : AUC0-12,
The area under the concentration-time curve from time zero (pre-dose) to 24 h post-dose, for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  The area under the concentration-time curve from time zero (pre-dose) to 24 h post-dose: AUC0-24,
The area under the concentration-time from time zero (pre-dose) to the time of last quantifiable concentration, for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  The area under the concentration-time from time zero (pre-dose) to the time of last quantifiable concentration: AUC0-t,
The apparent terminal elimination half-life, for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  The apparent terminal elimination half-life : t1/2,
Pre-morning dose concentration, for stiripentol relevant metabolites in plasma | Day 1 and Day 15 when applicable
  Pre-morning dose concentration : Cmin.
Total amount excreted over the time interval between 0 and 12 h, for stiripentol relevant metabolites in urine | Day 1 and Day 15 when applicable
  Total amount excreted over the time interval between 0 and 12 h : Ae0-12
Total amount excreted over the total time interval of urine collection i.e. ]0 - 24] h, for stiripentol relevant metabolites in urine | Day 1 and Day 15 when applicable
  Total amount excreted over the total time interval of urine collection i.e. ]0 - 24] h : Ae0-24
The fraction of the dose excreted in urine over the total time interval of urine collection i.e. ]0 - 24] h, for stiripentol relevant metabolites in urine | Day 1 and Day 15 when applicable
  The fraction of the dose excreted in urine over the total time interval of urine collection i.e. ]0 - 24] h : fe0-24
The renal clearance, for stiripentol relevant metabolites in urine | Day 1 and Day 15 when applicable
  The renal clearance : CLr

CONTACTS AND LOCATIONS:
Overall Officials: Diyan Genov, MD, Principal Investigator — Comac Medical
Locations (1):
- Mc Comac Medical, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No